CLINICAL TRIAL: NCT06790615
Title: To Compare Thread Technique Versus Aspiration Plus Steroid Injection of Wrist Ganglion in Terms of Frequency of Recurrence
Brief Title: Comparison of Thread Technique Versus Aspiration Plus Steroid Injection for Wrist Ganglion Recurrence
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Benazir Bhutto Hospital, Rawalpindi (Other Government)
Responsible Party: Principal Investigator, Fazal Hussain Shah, Consultant Surgeon, Benazir Bhutto Hospital, Rawalpindi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERC/19/15(b)
Record Dates: First submitted 2025-01-14; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Ganglion Cyst
Keywords: Cyst; ganglion; Thread technique; Wrist swelling
MeSH Terms: conditions — Ganglion Cysts; Cysts

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thread technique (Experimental): The thread technique was used for the wrist ganglion
  Interventions: Other: Silk suture
- Steriod injection (Active Comparator): Steriod injection was given into the cyst after aspiration
  Interventions: Drug: methyl prednisolone acetate

INTERVENTIONS:
Drug: methyl prednisolone acetate — methyl prednisolone acetate was injected after the aspiration
  Arms: Steriod injection
Other: Silk suture — The silk suture was used for threading technique
  Arms: Thread technique

SUMMARY:
This study is a randomized controlled trial comparing two treatment methods for wrist ganglion cysts to evaluate which method has a lower recurrence rate. Ganglion cysts are non-cancerous lumps commonly found on the wrist, arising from joint capsules or tendon sheaths. They are often painless but may cause discomfort or cosmetic concerns.

The primary objective of this study was to compare the recurrence rates of wrist ganglia treated with two methods:

Thread technique: Inserting a silk thread through the cyst to allow drainage. Aspiration plus steroid injection: Removing the cyst fluid with a needle followed by injecting a corticosteroid to reduce inflammation.

Study Design The trial was conducted at HIT Hospital, Taxila, from June to December 2020. It included 60 participants aged 18-50 years, divided equally into two groups. Group A underwent the thread technique, and Group B received aspiration and steroid injections. Patients were followed up at intervals of 2 weeks, 6 weeks, 3 months, and 6 months to monitor for cyst recurrence.

Methods Thread Technique: A silk suture was passed through the cyst, allowing its contents to drain. Patients were instructed to massage the area daily for one week. The thread was removed once drainage ceased.

Aspiration and Steroid Injection: Fluid was removed using a needle, and 40 mg of methylprednisolone acetate was injected into the cyst cavity.

Both procedures were performed under local anesthesia in an outpatient setting.

DETAILED DESCRIPTION:
INTRODUCTION Ganglia is the commonest cause of referral for upper extremity soft tissue tumors. More than 50% of referrals belong to this category. Ganglion originated from joint capsule or tendon sheaths. The most common site is wrist followed by the vicinity of interphalangeal joints. The dorsal ganglia mostly originate from scapho-lunate interosseous ligament while volar may arise from radio-scaphoid joint or scapho-trapezial joint. The most common presentation is painless lump at abovementioned areas. The pain may arise when the ganglia exert pressure effects during movements. The diagnosis is clinical in most cases and additional laboratory, or radiological investigations are often not helpful.

The treatment of ganglia is mainly sought out due to pain or cosmetic reasons. Management is tailored accordingly ranging from simple reassurance to surgical excision with in between options of aspiration with and without steroid injection, hyaluronidase injection and thread or seton insertion. The surgical excision may be orthoscopic as well. The aspiration and steroid injection may be cost effective but is associated with skin pigmentation, atrophic changes, and increased chances of recurrence. Surgical excision is associated with operative cost, infections and possible chances of nerve, tendon, or joint damage. The thread technique has been seen in some early research but to some extent has been ignored irrespective of the fact that it is cost effective and has comparable outcomes. The recurrence is common with all the current procedures.

Investigators conducted this study to determine the frequency of recurrence of wrist ganglia between threading technique and aspiration plus steroid injection. Both these procedures are being practiced as outpatient procedures in our setup. There is paucity in local and international literature regarding this specific subject. The result of our study would provide us with better insight into this subject and will leave us with a better choice to treat wrist ganglia..

METHODS AND MATERIALS This randomized controlled trial was conducted at HIT hospital Taxila from January 2020 to June 2020 for period of one year with clinical diagnosis of wrist ganglion. This study was conducted in accordance with ethical standards and principles. Institutional Review Board (IRB) or Ethics Committee approval was obtained prior to the commencement of the research (Reference number: ERC/19/15(b). Informed consent was acquired from all participants involved in the study. The research was conducted with respect for participant privacy, confidentiality, and autonomy. The sample size of 60 patients (30 in each group) was calculated by taking recurrence rates of 4% and 43% for threading technique and aspiration plus steroid injection respectively from a study.9 The level of significance was 5% and power of test was 90%. Randomization of patients was done into two equal groups by computer generated numbers. In group A, the aspiration of ganglion was done by 18G needle attached to a 10 ml syringe. After full aspiration, methylprednisolone (40 mg/ml) was injected into the cavity. In group B, the silk suture size 1 was passed horizontally through the ganglion and tied over sterile gauze. The evacuation of mucinous contents was done manually, and patients were instructed to do manual massage three times daily for 7 days. The thread was removed after 2 weeks or when only serosanguinous discharge was observed at the entry points of thread. Both procedures were done with full aseptic measures and under local anesthesia of 1% lignocaine. The patients were followed in OPD after 2 weeks, 6 weeks, 3 months, and 6 months. The recurrence was noted down on specially designed proforma for study.

The data was analyzed by Statistical Package for Social Science (SPSS) version 25 registered for Microsoft windows. The quantitative variables like age and duration of disease were expressed by mean and standard deviation. The qualitative variables like gender and recurrence at follow up visits were expressed as frequency and proportions. Both groups A and B were compared among each other in terms of recurrence at 2 week, 6 weeks, 3 months, and 6 months by Chi Square test. P value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical and radiological diagnosis of wrist ganglion.
* Both genders.
* Age range of 18 to 50 years.

Exclusion Criteria:

* Patients with a history of previous invasive treatments.
* Patients with compound ganglion.
* Patients with diabetes mellitus.
* Patients with bleeding diathesis. Patients with immunosuppression. Patients with rheumatoid arthritis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence | 2 weeks
  Number of patients with recurrence of ganglion cyst
Recurrence | 6 weeks
  Number of patients with recurrence of ganglion cyst
Recurrence | 3 months
  Number of patients with recurrence of ganglion cyst
Recurrence | 6 months
  Number of patients with recurrence of ganglion cyst

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Basit, MBBS, FCPS, Principal Investigator — POF Hospital, Wah Cantt.
Locations (1):
- PAF Hospital, Islamabad, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT06790615/Prot_SAP_ICF_000.pdf